CLINICAL TRIAL: NCT00841373
Title: Ranibizumab Supplementing Panretinal Photocoagulation as Treatment for Iris/Angle Neovascularization in Retinal Ischemic Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Southern New England Retina Associates (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Mary Savell, Madgalena G. Krzystolik, M.D., Southern New England Retina Associates
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100,611
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Retinal Ischemia
Keywords: Retinal ischemia: Iris/Angle Neovascularization
MeSH Terms: interventions — Lasers; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Panretinal Photocoagulation
  Interventions: Procedure: Panretinal Photocoagulation
- 2 (Active Comparator): Ranibizumab Supplementing Panretinal Laser Photocoagulation
  Interventions: Procedure: Panretinal Photocoagulation and intravitreal injection of ranibizumab

INTERVENTIONS:
Procedure: Panretinal Photocoagulation — Panretinal Photocoagulation treatment
  Arms: 1
Procedure: Panretinal Photocoagulation and intravitreal injection of ranibizumab — Panretinal photocoagulation and ranibizumab
  Other Names: laser and Lucentis
  Arms: 2

SUMMARY:
The object of the study is to compare treatment of iris/angle neovascularization with panretinal photocoagulation (laser) to treatment with panretinal photocoagulation and an anti-angiogenic drug: ranibizumab.

DETAILED DESCRIPTION:
A.To obtain preliminary data on the safety and tolerability of ranibizumab (0.5 mg)in patients with new or progressive neovascularization of the iris or angle due to retinal ischemic diseases in addition to treatment with PRP using the incidence and severity of adverse events identified by subjenc reporting vital signs, and ocular examition.

B.To assess the proportion of patients who fail to experience regression of iris and angle neovascularization documented by the clinical examination, iris florescein angiography and gonioscopic evaluation.

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet the following criteria to be eligible for study entry:

1. Signed informed consent and authorization of use and disclosure of protected health information
2. Age = 18 years
3. Presence of iris neovascularization and or angle neovascularization due to any retinal ischemic disease that is new onset or noted to progress recently on the slit lamp examination or gonioscopy
4. Best corrected visual acuity in the study eye 20/20 (Snellen equivalent using EDTRS protocol at 4 meters) to light perception. Only one eye will be enrolled in the study. If both eyes are eligible, the investigator will select the eye to be enrolled. Visual acuity in the non-study eye must be better than no light perception
5. Patient is able and willing to return for all scheduled visits

Exclusion Criteria:

1. Use of intraocular or periocular injection of steroids (for, example triamcinolone) in the study eye within 3 months of the study
2. Use of intraocular injection of anti-angiogenic drugs in the study eye and or participation in a clinical trial using an antiangiogenic treatment within 45 days from the enrollment in the study.
3. Acute endophthalmitis within 1 month.
4. Recent rhegmatogenous retinal detachment or macular hole surgery within last 2 months
5. Uncontrolled uveitis in the last month.
6. Treatment with PRP within 2 weeks of the study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of adverse events identified by subject reporting, vital signs, and ocular exam. | 1 to 12 months
The proportion of patients who fail to maintain regression of iris and angle neovascularization documented by the clinical examination iris fluorescein angiography and gonioscopic evaluation. | 1 to 12 months

SECONDARY OUTCOMES:
The mean change in best corrected visual acuity score | 1 to 12 months
The percentage/number of patients that experience vision loss of 30 letters or less | 1 to 12 months
The percentage number of patients that experience vision improvement of more than 15 letters | 1 to 12 months
The percentage/number of patients whose vision progressed to no light perception | 1 to 12 months
The mean change in macular thickness on OCT | 1 to 12 months
The percentage/number of eyes that will require surgical intervention to maintain the intraocular pressure or useful vision | 1 to 12 months
The percentage/ number of eyes that will require anti-glaucoma medications to control intraocular pressure | 1 to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena G Krzystolik, MD, Principal Investigator — Southern New England Retina Associates
Locations (1):
- Southern New England Retina Associates, Providence, Rhode Island, United States